CLINICAL TRIAL: NCT00010478
Title: Acupuncture and Hypertension-Efficacy and Mechanisms
Brief Title: Acupuncture and Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT000129-02 (NIH); NCT00008905 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
Although traditional Chinese medicine advocates the use of acupuncture not only to induce analgesia but also to treat essential hypertension, acupuncture's postulated antihypertensive efficacy in humans has not been subjected to rigorous Western scientific testing. Before advocating acupuncture as an effective complementary/alternative medicine strategy for essential hypertension, it is necessary to demonstrate that the beneficial effects of acupuncture are scientifically robust, long-lasting, and explicable in terms of modern scientific mechanisms. In spontaneously hypertensive rats, acupuncture-like electrical stimulation of thinly myelinated (Group III) somatic afferents activates central endorphin (naloxone-sensitive) pathways that elicit long-lasting decreases in sympathetic nerve activity (SNA) and blood pressure. The ability to record SNA with microelectrodes in conscious humans provides a new opportunity to test this novel mechanistic hypothesis in patients undergoing electroacupuncture, a modification of the ancient technique that provides a quantifiable and reproducible stimulus to human skeletal muscle afferents. Using a randomized, double-blind placebo-controlled design, we will test the following major hypotheses: Electroacupuncture produces a long-lasting reduction in SNA, thereby providing a safe and effective complementary treatment of human hypertension. Given the enormous interest in acupuncture by our lay public, but the paucity of Western scientific data about its efficacy in cardiovascular disorders, our studies in normotensive and hypertensive humans should provide a conceptual framework for deciding whether to accept or reject the large body of Chinese (and Russian) literature advocating acupuncture as a safe and effective treatment of essential hypertension and other cardiovascular disorders (such as heart failure, and myocardial ischemia).

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal blood pressures or blood pressures over 120/80 up to 165/105

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern, Dallas, Texas, United States